CLINICAL TRIAL: NCT00685490
Title: Vitrectomy for Persistent Macular Edema in Branch Retinal Vein Occlusion
Brief Title: Vitrectomy for Branch Retinal Vein Occlusion
Status: Completed | Type: Observational
Sponsor: Shinjo Ophthalmologic Institute (Other)
Responsible Party: Kazuyuki Kumagai, Shinjo Ophthalmologic Institute
Other Study IDs: KK-R-207-430R1; Kumagai BRVO
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Vitrectomy
Keywords: branch retinal vein occlusion; internal limiting membrane; macular edema; vitrectomy
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Surgical: Retrospective chart review of 70 eyes of 70 consecutive patients who underwent PPV, with and without ILM peeling, for persistent macular edema associated with BRVO
  Interventions: Procedure: Vitrectomy w/o ILM peeling for macular edema with BRVO

INTERVENTIONS:
Procedure: Vitrectomy w/o ILM peeling for macular edema with BRVO — Concurrent phacoemulsification and intraocular lens insertion in the capsular bag was performed, followed by PPV with separation of the posterior hyaloid from the optic disk and posterior retina with a posterior vitreous detachment was not present. Indocyanine green (ICG)-assisted peeling was performed in all consecutive patients between April 2000 and June 2003. 0.1% ICG solution was injected over the macular region. Immediately after application, the dye was washed out using a vitreous cutter. Repeated injection of ICG was not required. Triamcinolone acetonide (TA)-assisted ILM peeling was performed in all consecutive patients from July 2003 to November 2006.

SUMMARY:
To evaluate the long term outcomes of pars plana vitrectomy (PPV), with and without internal limiting membrane (ILM) peeling, in eyes with persistent macular edema secondary to branch retinal vein occlusion (BRVO).

Results suggest the following hypothesis:

* PPV, with and without ILM peeling, appears to be beneficial in eyes with persistent macular edema due to BRVO
* Effectiveness is maintained long term
* ILM peeling does not significantly affect postoperative best corrected visual acuity (BCVA)

ELIGIBILITY:
Inclusion Criteria:

* duration of symptoms lasting 27 weeks

Exclusion Criteria:

* vitreous hemorrhage
* severe cataract
* biomicroscopic vitreomacular traction and epiretinal membrane
* previous vitreoretinal surgery
* other ocular diseases that could contribute to visual loss.
* patients with macular branch vein occlusion
* patients with a history of previous grid laser photocoagulation

Ages: 45 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 consecutive patients who underwent PPV, with and without OLM peeling, for persistent macular edema associted with BRVO
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 1995-07; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Reporting of the long term outcomes of PPV, with and without ILM peeling, in eyes with persistent macular edema secondary to BRVO | 11 years

SECONDARY OUTCOMES:
Elevate the effectiveness of ILM peeling | 11 years

CONTACTS AND LOCATIONS:
Overall Officials: Kazuyuki Kumagai, MD, Principal Investigator — Shinjo Ophthalmologic Institute
Locations (1):
- Shinjo Ophthalmologic Institute, Miyazaki, Miyazaki, Japan